CLINICAL TRIAL: NCT00041691
Title: A Phase I, Single Dose Escalating Study to Investigate the Tolerability, Pharmacokinetics and Dosimetry of 90 Y-Humanized MN-14 IgG in Colorectal Cancer Patients With Limited Residual Disease After Primary or Salvage Surgery
Brief Title: Safety Study of 90Y-hMN14 to Treat Colorectal Cancer Patients With Limited Residual Disease After Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-hMN14-06
Record Dates: First submitted 2002-07-12; First posted 2002-07-15 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2003-01

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Cancer; Colon Cancer; Rectal Cancer; Colorectal Neoplasms; Colorectal Carcinoma; Colorectal Tumor
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — labetuzumab

INTERVENTIONS:
Drug: hMN14 (labetuzumab)

SUMMARY:
The purpose of this trial is to determine the safety of 90Y-hMN14 at different dose levels in the treatment of residual colorectal cancer following recent surgery.

ELIGIBILITY:
Disease Characteristics:

* Patients with documented histologic and cytologic diagnosis of colon or rectal malignancy
* Patients with documented status post surgical resection of primary cancer or metastases
* Limited residual disease (i.e., CEA serum levels < 15 ng/mL and negative baseline CT scans, or no lesion > 1 cm)

Prior/Concurrent Therapy:

* Patients must have completed chemotherapeutic agents, biologic therapy, radiotherapy, other investigational therapy for cancer, or surgical procedures at least six weeks prior to study entry.
* Patients must have recuperated from surgery and toxicities (as a result of previous therapy) sufficiently prior to study entry
* Biologic Therapy: Patients who have received a murine, chimeric, CDR-grafted (humanized), or human IgG will be eligible provided pre-study evaluations demonstrate no significant reactivity with hMN-14 IgG (i.e., HAHA)
* Radiotherapy: No prior external beam irradiation to a field that includes more than 30% of the red marrow. No prior radiation to maximal tolerable levels for any critical organs (e.g., 3000 cGy for the liver; 2000 cGy for the lungs and kidneys)

Patient Characteristics/Inclusion Criteria:

* Performance Status: Patients with Karnofsky performance status > 70%
* Hematopoietic: ANC >/= 1.5 x 10/L; Hemoglobin >/= 10 g/dL; Platelets >/= 100 x 10/L
* Renal: Serum Creatinine </= 1.5 x ULN
* Hepatic: Serum Bilirubin </= 1.5 ULN; AST and ALT </= 2.5 x ULN; Alk Phosphatase </= 2.5 x ULN
* Cardiovascular: Patients with LVEF >/= 50% by required MUGA/2D-ECHO tests
* Pulmonary: Patients with DF and FEV1 >/= 60% by required Pulmonary Function Tests
* Central Nervous System: Patients with known metastatic disease to the CNS are excluded.
* Other: Patients agreeing to use a medically effective method of contraception during and for a period of three months after the treatment period. A pregnancy test will be preformed on each premenopausal female of childbearing potential immediately prior to entry into study. Patients must understand and give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Overall Officials: Lauri Welles, MD, Study Chair — Gilead Sciences; Terence Rugg, MD, Study Director — Gilead Sciences
Locations (2):
- United States (2):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Virginia Mason Medical Center, Seattle, Washington